CLINICAL TRIAL: NCT05644509
Title: A Clinical Pharmacological Study of Intravenous Administration of Vesicular Stomatitis Oncolytic Virus Injection (Revottack）Combined PD-1 Inhibitor in Patients With Advanced Malignant Solid Tumor
Brief Title: Study on the Treatment of Advanced Malignant Solid Tumor With Revottack and PD-1 Inhibitor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LWY22078CXY
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Tumor
Keywords: Oncolytic Virus; Revottack; PD-1(Toripalimab); Intravenous Injection; immunotherapy; immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncolytic Virus Injection（Revottack）+PD-1 (Experimental): In the first three cycles, the subjects were administered on the first day and the sixth day of each cycle respectively; At the beginning of the fourth cycle, the subjects were administered on the sixth day of each cycle, 14 days a cycle.
  PD-1 inhibitor(Toripalimab) Intravenous infusion, once every 2 weeks from the 6th day.
  Interventions: Biological: Oncolytic Virus Injection（Revottack）+PD-1

INTERVENTIONS:
Biological: Oncolytic Virus Injection（Revottack）+PD-1 — Intravenous injection of Revottack injection combined with PD-1(Toripalimab） inhibitor

SUMMARY:
This is a one arm, open clinical pharmacological exploration study initiated by researchers to evaluate the safety and effectiveness of vesicular stomatitis oncolytic virus injection (Revottack) combined with PD-1 inhibitor in patients with advanced malignant solid tumors.

The purpose of this study is to evaluate the safety, tolerability, anti-tumor activity, immunogenicity, immune response, pharmacokinetic (PK) characteristics and shedding characteristics of Revottack injection combined with PD-1 inhibitor in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a one arm, open clinical pharmacological exploration study initiated by researchers to evaluate the safety and effectiveness of vesicular stomatitis oncolytic virus injection (Revottack) combined with PD-1 inhibitor in patients with advanced malignant solid tumors.

This study is planned to enroll 6-10 patients with advanced solid tumors. Subjects will receive the administration of revottack and PD-1( Toripalimab)inhibitor at a given time.

The purpose of this study is to evaluate the safety, tolerability, anti-tumor activity, immunogenicity, immune response, pharmacokinetic (PK) characteristics and shedding characteristics of Revottack injection combined with PD-1 inhibitor in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* The age at the time of signing the informed consent is ≥ 18 years old, regardless of gender;
* Patients with advanced malignant solid tumor confirmed by histology or cytology; Failure in standard treatment (disease progression or intolerable treatment after treatment) and no effective treatment means, or no standard treatment scheme, or inability to obtain standard treatment due to objective conditions.
* According to RECIST 1.1, there is at least one assessable tumor focus with the longest diameter ≥ 10mm (if it is a malignant lymph node, the short diameter ≥ 15mm is required);
* ECOG physical strength score 0-2;
* Full organ function:

Blood system (no blood transfusion or hematopoietic stimulator treatment within 14 days) Absolute neutrophil count (ANC) ≥ 1.5 × 109/L Platelet (PLT) ≥ 75 × 109/L Hemoglobin (Hb) ≥ 80g/L Lymphocyte absolute value (LYM) ≥ 0.8 × 109/L liver function Total bilirubin (TBIL) ≤ 1.5 × ULN Alanine aminotransferase (ALT) ≤ 3 × ULN (Patients with liver metastasis or liver cancer: ≤ 5 × ULN ) Aspartate aminotransferase (AST) ≤ 3 × ULN (Patients with liver metastasis or liver cancer: ≤ 5 × ULN) renal function Creatinine clearance rate (Ccr) > 50ml/min/1.73m2 (calculated according to Cockcroft Gault formula) Coagulation function test Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN International normalized ratio (INR) ≤ 1.5 × ULN

* Eligible patients (male and female) with fertility must agree to work in Revottack Use reliable contraceptive methods (hormone or barrier method or abstinence) within 6 months after injection; The blood pregnancy test of female patients of childbearing age must be negative within 7 days before enrollment;
* Subjects must give informed consent to the study before the study, and voluntarily sign a written informed consent form.

Exclusion Criteria:

* Patients with active CNS metastasis and/or carcinomatous meningitis are known or found during screening. However, the following subjects are allowed to be included in the group: ① Patients with asymptomatic brain metastasis (that is, patients without progressive central nervous system symptoms caused by brain metastasis do not need to use corticosteroids) can participate. ② Subjects who had been treated and had stable brain metastases for at least 2 months had no evidence of new or expanded brain metastases.
* He received chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor treatments within 2 weeks before the first use of the study drug;
* Participated in other unlisted clinical studies within 4 weeks before the first use of the study drug;
* Major organ surgery (excluding puncture biopsy) or significant trauma occurred within 4 weeks before the first use of the study drug, or major elective surgery required during the study period.
* Patients who received systemic corticosteroids (prednisone>10mg/day or equivalent dose of the same drug) or other immunosuppressants within 14 days before the first use of the study drug; The following cases are excluded: local, eye, intra articular and intranasal corticosteroids are used for treatment; Short term use of corticosteroids for prevention and treatment;
* Have received other oncolytic virus treatment within 8 weeks before the first use of the study drug;
* Any vaccine was inoculated within 7 days before the first use of the study drug;
* Antiviral drugs were used within 2 weeks before the first use of the study drug, and long-acting interferon was used within 4 weeks;
* The adverse reaction of previous anti-tumor treatment has not recovered to ≤ 1 level (except for the toxicity judged by the researcher as no safety risk, such as alopecia, hypothyroidism stabilized by hormone replacement therapy, etc.);
* Uncontrolled active infection exists, which may seriously affect the efficacy and safety evaluation as judged by the researcher;
* Have a history of immunodeficiency, including HIV antibody test positive;
* Active hepatitis B (HBsAg positive and HBV DNA>the lower detection limit of the research center), or hepatitis C virus infection (anti HCV positive or HCV RNA positive), or syphilis infection;
* Cardiovascular and cerebrovascular diseases shall conform to any of the following:

  1. Poor control of hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg);
  2. Cardiac function ≥ Grade 2 congestive heart failure (NYHA classification);
  3. Arrhythmias requiring clinical intervention (including QTc ≥ 450ms (male) and QTc ≥ 470ms (female));
  4. Serious arteriovenous thromboembolism events, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis or any other serious thromboembolism;
* The third space effusion that cannot be controlled clinically is not suitable to be included in the group according to the judgment of the researcher;
* Patients with active or ever suffered from autoimmune diseases that may recur (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except patients with clinically stable autoimmune thyroiditis;
* Known alcohol or drug dependence;
* Mental disorders or poor compliance;
* Pregnant or lactating women;
* The investigator believes that the subject is not suitable to participate in this clinical study because of other serious systemic diseases or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  Graded according to the NCI CTCAE version 5.0.
Objective response rate | Up to 2 years
  Assess the proportion of patients who achieved complete or partial response
Disease control rate | Up to 2 years
  Assess the proportion of patients who achieved complete or partial or stable response
The changes from baseline of lymphocyte counts | Up to 28 days
  The changes from baseline of Peripheral blood lymphocyte subtypes counts
The concentration of antiviral antibody | Up to 22 Weeks
  The concentration of antiviral antibody of Revottack in blood
The rate of subjects with viral shedding of Revottack | Up to 22 Weeks
  The rate of subjects with viral RNA in the secretion
The Tmax of Viral RNA in blood | Up to 22 Weeks
  Time to peak viral RNA concentration
The Cmax of Viral RNA in blood | Up to 22 Weeks
  The peak viral RNA concentration

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No